CLINICAL TRIAL: NCT06527729
Title: Sildenafil-loaded Lipid-based Nanocarrier as a Potential Therapy for Alopecia Areata: A Randomized Clinical Study
Brief Title: A Novel Formulation of Sildenafil-loaded Nanocarriers for Treatment of Alopecia Areata
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Fathy Ahmed, Lecturer of Dermatology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sildenafil-loaded nanocarriers
Record Dates: First submitted 2024-07-14; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to use either topical 5% minoxidil gel or topical 1% sildenafil-loaded liposomes twice daily for a period of 8 weeks.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Topical 5% minoxidil gel was applied twice daily for a period of 8 weeks.
  Interventions: Drug: minoxidil gel
- Group 2 (Experimental): Topical 1% sildenafil-loaded liposomes was applied twice daily for a period of 8 weeks.
  Interventions: Drug: sildenafil-loaded liposomes

INTERVENTIONS:
Drug: sildenafil-loaded liposomes — Topical 1% sildenafil-loaded liposomes was applied twice daily for a period of 8 weeks over patchy alopecia areata of the scalp.
  Arms: Group 2
Drug: minoxidil gel — Topical 5% minoxidil gel was applied twice daily for a period of 8 weeks.
  Arms: Group 1

SUMMARY:
Alopecia areata (AA) is a common cause of nonscarring alopecia that occurs in a patchy, confluent, or diffuse pattern. Many theories were implicated in pathogenesis of AA, such as an autoimmune lymphocytic attack of the hair, genetic basis, and environmental factors. Clinically, AA presents as a well-circumscribed patch of sudden hair loss. It affects any hair bearing area with the scalp being the most commonly affected site .

Dermoscopy is a noninvasive technique for the clinical diagnosis of many skin diseases. Dermoscopy is now considered as a valuable tool in diagnosis of variable skin lesions. Scalp dermoscopy (Trichoscopy) does not only facilitate diagnosis of hair disorders but also give clues about disease stage and progression.

The most common trichoscopic features of AA are yellow dots, micro-exclamation mark hairs, tapered hairs, black dots, broken hairs, and regrowing upright or regrowing coiled hairs. Trichoscopic characteristics have a clinical significance in AA for diagnosis and prognosis.

The treatment of alopecia areata involves promotion of hair growth (for instance with topical minoxidil application), immunosuppression (intralesional or systemic steroid therapy, phototherapy) or immunomodulation (anthralin, dinitrochlorobenzene, diphenylcyclopropenone, squaric acid dibutylester).Unfortunately, there is currently no cure for this chronic disease, and despite the presence of a wide variety of therapeutic options, none is universally proven to induce and/or sustain remission. Development of new drugs and formulations is urgently needed

Sildenafil, a phosphodiesterase 5 (PDE5) inhibitor, is known to increase the intracellular level of cyclic guanosine monophosphate (cGMP), which causes vasodilation. Sildenafil was first approved in 1998 for erectile dysfunction, but since then additional uses for the drug have been found. A previous study demonstrated the significant therapeutic potential of sildenafil on hair growth and proposed its potential use in treatment of alopecia. It has been shown that it enhances proliferation of human dermal papilla cells (hDPCs) and up-regulates the mRNA expression of vascular endothelial growth factor (VEGF) and platelet-derived growth factor (PDGF), which are responsible for hair growth. Additionally, sildenafil up-regulates the levels of phosphorylated ERK and accelerates anagen induction by stimulating perifollicular vessel formation after topical application in mice.

DETAILED DESCRIPTION:
The aim of the present work was to optimize sildenafil-loaded liposomes which could enhance percutaneous absorption and follicular penetration of sildenafil achieving improved therapeutic efficiency with minimal unnecessary side effects due to oral administration.

In addition, the study aimed to assess the efficacy of topical sildenafil-loaded liposomes formulation compared with topical minoxidil therapy for the treatment of patchy AA of the scalp through examination of its clinical effects along with dermoscopic findings.

Materials Lipoid S75 (phosphatidylcholine (70 %) with fat-free soybean phospholipids) was kindly donated by lipoid company (Germany). Sildenafil citrate was purchased from Fagron Iberica SAU. Acetonitrile HPLC reagent was purchased from Fisher Chemical. Ultrapure water was. Cholesterol was purchased from Fluka chemical co. (India). Ethanol (absolute) was purchased from El-Nasr Pharmaceuticals, (Egypt). All reagents and chemicals were purchased from (Sigma Aldrich).

Methodology Preparation of SIL-LIP using spraying technique SIL-LIP were formulated using spraying method. Pre-calculated amounts of Lipoid s75, cholesterol and sildenafil were dissolved in 2 ml of absolute ethanol and the prepared solution was transferred to a spraying apparatus [20]. In a closed system, the alcoholic solution of sildenafil and lipids was sprayed (100 ul were sprayed every 10 seconds) onto the surface of 2 ml distilled water containing sucrose (9% w/v) with stirring at 1250 rpm at 25º C. Stirring was maintained until complete evaporation of ethanol. To guarantee complete annealing of the formed liposomes, SIL-LIP were kept at 4°C overnight [21]. SIL-LIP were imaged using (JEM-1400,-Jeol,-Tokyo,-Japan) maintained at 80-kV. SIL-LIP was-left for ten minutes at 25°C before examination on carbon-coated-copper-grid.

Particle size measurement To gain more insight into size and size distribution, laser light diffraction was employed. the Prepared SIL-LIP were diluted with deionized water and was analyzed with Mastersizer 3000E Malvern Instruments, UK at 25°C. The result was the average of three repeated values.

Entrapment efficiency (E.E) of prepared liposomes

The EE% was determined by centrifugation of liposomal suspension at 1.000 rpm for 45 min at 4 °C to isolate the unentrapped sildenafil in the supernatant for indirect determination of EE% . The amount of sildenafil in the supernatant was determined by UV spectrophotometer (Spectronic Genesys®, Winspec Software, Spectronic, USA) at 228 nm . EE (%) was calculated as follows:

EE (%) = [(Qi -Qs)/Qt] × 100 where Qi is the initial amount of the sildenafil added during preparation and Qs is the sildenafil amount determined in the supernatant after centrifugation Clinical study A prospective randomized controlled study was conducted in the department of Dermatology, Assiut University Hospital including patients with patchy AA of scalp, aged between 10 and 40 years. Patients having alopecia totalis/universalis, or ophiasis, those with systemic and/or other dermatological diseases and those receiving treatment for AA in the previous 3 months were excluded.

This study was conducted in compliance with the guidelines of the Declaration of Helsinki and the study protocol was approved by the Research Ethics Committee of Faculty of Medicine, Assiut University (IRB no. 17300458). Informed consent was obtained from all patients before enrolments.

At the initial visit, full history taking and thorough clinical examination was done for all patients. The diagnosis was established based on both clinical and dermoscopic examination.

Treatment Protocol

Patients were randomly assigned to use either topical 5% minoxidil gel or topical 1% sildenafil-loaded liposomes twice daily for a period of 8 weeks.

Assessment criteria

Clinical evaluation was performed by the comparison of serial photographs of the lesions to the baseline ones. Severity of Alopecia Tool (SALT) score was calculated, at baseline, 4 weeks and 8 weeks and the average percentage of hair re-growth was determined using the SALT scoring system for hair re-growth and graded as A0: no change or further hair loss, A1: 1-24% hair re-growth, A2: 25-49% hair re-growth, A3: 50-74% hair regrowth, A4: 75-99% hair re-growth, and A5: 100% hair re-growth .

Dermoscopic examination was carried out before treatment and at 4 and 8 weeks, using the handheld dermoscope (DermLite DL4, 3Gen, Inc., San Juan Capistrano, CA 92675). Baseline and post-therapy digital photographs of dermoscopic fields were taken using an iPhone 6S smartphone camera. Dermoscopic features of AA were evaluated including yellow dots, black dots, broken hair, exclamation-mark hairs, short vellus hair and regrowing hair . Two dermoscopic fields were examined; one from the center and the other at 3 o'clock position of the alopecia patch. Trichoscopic parameters in each field were evaluated and quantified.

Data analysis was done using the SPSS software version 24 (SPSS Inc., Chicago, IL, USA). The Chi-square test and Mann-Whitney test were used for comparison of qualitative data and quantitative data, respectively. P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

• Patients with a clinical and dermoscopic diagnosis of patchy alopecia areata of the scalp.

Exclusion Criteria:

* Alopecia totalis/universalis.
* Ophiasis.
* Those with systemic and/or other dermatological diseases.
* Those receiving treatment for a lopecia areata in the previous 3 months.

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
The efficacy of topical sildenafil-loaded liposomes formulation compared with topical minoxidil therapy for the treatment of patchy alopecia areata | 8 weeks
  the comparison of serial photographs of the lesions to the baseline ones. Severity of Alopecia Tool (SALT) score was calculated, at baseline, 4 weeks and 8 weeks and the average percentage of hair re-growth was determined using the SALT scoring system for hair re-growth and graded as A0: no change or further hair loss, A1: 1-24% hair re-growth, A2: 25-49% hair re-growth, A3: 50-74% hair regrowth, A4: 75-99% hair re-growth, and A5: 100% hair re-growth
Dermoscopic asessment | 8 weeks
  Dermoscopic examination was carried out before treatment and at 4 and 8 weeks, using the handheld dermoscope (DermLite DL4, 3Gen, Inc., San Juan Capistrano, CA 92675). Baseline and post-therapy digital photographs of dermoscopic fields were taken using an iPhone 6S smartphone camera. Dermoscopic features of AA were evaluated including yellow dots, black dots, broken hair, exclamation-mark hairs, short vellus hair and regrowing hair. Two dermoscopic fields were examined; one from the center and the other at 3 o'clock position of the alopecia patch. Trichoscopic parameters in each field were evaluated and quantified.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Fathy, MD, Principal Investigator — Assiut university, Faculty of Medicine, Egypt
Locations (1):
- Faculty of Medicine, Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Owis AI, El-Hawary MS, El Amir D, Refaat H, Alaaeldin E, Aly OM, Elrehany MA, Kamel MS. Flavonoids of Salvadora persica L. (meswak) and its liposomal formulation as a potential inhibitor of SARS-CoV-2. RSC Adv. 2021 Apr 12;11(22):13537-13544. doi: 10.1039/d1ra00142f. eCollection 2021 Apr 7. PMID 35423847